CLINICAL TRIAL: NCT04056143
Title: Development of Precision Medicine Platform for Pharmacogenomics of Novel Oral Anticoagulants (NOACs)
Brief Title: Precision Medicine Platform for Novel Oral Anticoagulants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Hsiang-Chun Lee, Assistant Professor, Kaohsiung Medical University
Other Study IDs: KMUHIRB-G(I)-20180026; 108-2622-B-037-003 -CC1 (Other Grant/Funding Number: Taiwan Ministry of Science and Technology)
Record Dates: First submitted 2019-07-30; First posted 2019-08-14 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Anticoagulant Adverse Reaction
Keywords: Thromboembolism; Oral anticoagulants; Adverse events; Pharmacogenomics; Precision Medicine
MeSH Terms: conditions — Thromboembolism | interventions — Pharmacogenomic Testing; Prothrombin Time; Partial Thromboplastin Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

GROUPS / COHORTS (4):
- Dabigatran: Subjects who are receiving long-term Dabigatran for certain clinical conditions, and without any contraindication are enrolled for this cohort group.
  Interventions: Diagnostic Test: Pharmacogenomics
- Rivaroxaban: Subjects who are receiving long-term Rivaroxaban for certain clinical conditions, and without any contraindication are enrolled for this cohort group.
  Interventions: Diagnostic Test: Pharmacogenomics
- Apixaban: Subjects who are receiving long-term Apixaban for certain clinical conditions, and without any contraindication are enrolled for this cohort group.
  Interventions: Diagnostic Test: Pharmacogenomics
- Edoxaban: Subjects who are receiving long-term Edoxaban for certain clinical conditions, and without any contraindication are enrolled for this cohort group.
  Interventions: Diagnostic Test: Pharmacogenomics

INTERVENTIONS:
Diagnostic Test: Pharmacogenomics — Subjects enrolled in this study are providing blood samples for completing a set of laboratory testing and pharmacogenomic analyses. They are requested to comply a Pharmacist interview and complete of assisted questionnaires.
  Other Names: Prothrombin time (PT), activated partial thromboplastin time (aPTT), Ecarin-based assay (for dabigatran), chromogenic anti-Xa assays (for rivaroxaban, apixaban, and edoxaban)

SUMMARY:
The anticoagulants have been developed with new generation for FDA-approved indications including treatment and prevention of venous, pulmonary, and systemic thromboembolism. While the prescription of new oral anticoagulants (NOAC) has increasingly and largely replaced warfarin in accordance of better efficacy and safety, there are still adverse effects, including incidental minor and major bleeding, and inefficacy in thrombosis prevention. The overarching goal of this study is to develop a Pharmacogenomics Platform that is specifically designed for NOACs, in order to optimize and personalize the prescription and to facilitate the precision medicine.

DETAILED DESCRIPTION:
Pharmaceutical companies have developed new oral anticoagulants (NOACs) to replace warfarin for prevention of systemic thrombo-embolization and embolic stroke in patients with atrial fibrillation or other thromboembolism diseases. The sale of NOACs has been increasing globally as the prevalence of atrial fibrillation increases in countries with aging population. Patients with high thromboembolism risk are also at high risk for major bleeding. The conservative strategy is not good for that more patients on reduced dose of NOACs had stroke. The clinical dilemma is how to justify the efficacy of NOACs in stroke prevention without encountering the incidental major bleeding from side effects. In order to solve this dilemma, the comprehensive evaluation of risk for thromboembolism, risk of bleeding, and genetic background on related to drug pharmacokinetics and response is essential. The primary goal of this project is to combine the clinical data and genetic information to develop a drug response evaluation platform to facilitate personalized and precision medicine for NOACs prescription.

Pharmacogenomics elucidates the drug response and side effect on the basis of individual genetic background. This proposed project will enroll clinical patients who have atrial fibrillation and indications for the prescription of NOACs. The information will be collected for clinical demographics, medical history of embolic stroke, thromboembolism events, any bleeding events, and concurrent use of other medicines. Peak level of NOAC in use, and post-drug coagulation test will be performed. The above data will be integrated for the pharmacogenomic analysis with multiple genes (CES1, ABCB1, SLCO1B1, CYP2C9*2, CYP2C9*3, VKORC, CYP3A4, MMP-9, ALOX5AP, MTHFR, FGB and eNOs). The single nucleotide polymorphism (SNPs) of gene clusters will be derived from this clinical study. These output results will be used to optimize the gene-array product that is specifically-designed for NOACs prescription.

The NOACs-specific gene-array for a precision prescription will be developed to help physicians to choose the right NOAC and the best dose for individualized patients. This tool will maximize thromboembolism prevention from the NOACs prescription along with the minimization of NOACs side effects. The product will be commercialized with great potential for the global market.

ELIGIBILITY:
Inclusion Criteria:

* Long-term indication for use of dabigatran
* Long-term indication for use of rivaroxaban
* Long-term indication for use of apixaban
* Long-term indication for use of edoxaban

Exclusion Criteria:

* Any contraindication for use of anticoagulants
* Prisoners
* pregnancy
* mental disorders
* history of any mechanical or prosthetic valve replacement
* hemodialysis or other renal replacement therapy
* congenital coagulation abnormalities
* autoimmune diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have one of the indications to use long-term anticoagulants, including atrial fibrillation, deep venous thrombosis, and pulmonary embolism.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of major bleeding events during any NOAC treatment | From date of enrollment until the date of first major bleeding events of any type or date of death, whichever came first, assessed up to 36 months.
  Any gastrointestinal, retroperitoneal, urinary tract, abnormal uterine bleeding, intracranial, intra-ocular or intra-spinal bleeding events that are noted in medical records or examination reports, or demonstrated by images studies including a computer tomography scan or a magnetic resonance imaging, or a sonography or an ophthalmoscope; or bleeding requiring surgery; or transfusion of ≥ 2 units (i.e. ≥ 500 mL) of packed red blood cells) or associated with a decrease in hemoglobin of ≥ 2.0 g/L episodes.
Number of minor bleeding events during any NOAC treatment | From date of enrollment until the date of first major bleeding events of any type or date of death, whichever came first, assessed up to 36 months.
  Any gastrointestinal, urinary tract, abnormal uterine, soft tissue, skin, conjunctival, nasopharyngeal, oral cavity bleeding events that are noted in medical records or examination reports, or demonstrated by images studies including an endoscopic examination, or a sonography or an ophthalmoscope; or requirement of blood transfusion of < 2 units (i.e. less than 500 mL) of packed red blood cells or associated with a decrease in hemoglobin of < 2.0 g/L episodes.
Number of thromboembolism events during any NOAC treatment | From date of enrollment until the date of first thromboembolism events of any type or date of death, whichever came first, assessed up to 36 months.
  Any clinical evident events of venous, pulmonary, or systemic thromboembolism that are noted in medical records or examination records, or demonstrated by images of an angiography, or a sonography, or a computer tomography scan, or an isotope phlebography.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Chun Lee, MD, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan